CLINICAL TRIAL: NCT04518943
Title: Multiphase Optimization Trial of Incentives for Veterans to Encourage Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-450
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Behavior; Exercise; Walking; Motivation; Hypertension; Depression; Body Mass Index
Keywords: sedentary behavior; walking; motivation
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Hypertension; Depression | interventions — Walking

STUDY DESIGN:
Intervention Model Description: The MOST trial design involves optimizing an intervention before it is tested against a usual control. It is optimized in that the various components of the intervention are tested against one another in a screening phase to assess which components add value to the intervention, and then only the valuable components are included in the final intervention. It is especially useful when an intervention has many potential combinations of components, as is the case with incentives. In a traditional trial, researchers would use theory or evidence from prior studies to choose an incentive design and test this package against usual care. Even if this package outperforms usual care in a randomized trial, the investigators cannot tell whether it was optimal. Some components could have provided no benefit or delivered in too small a dose to be effective. Other components could have been detrimental to subjects. There is no way to know if the components are all tested as a single package.
Who Masked: Investigator
Masking Description: Data will be masked to the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- F1M1P1R1 (Experimental): Financial Reward, mixed lottery, pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking
- N1M1P1R1 (Experimental): Non-financial reward, mixed lottery, pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking
- N1M1P1R0 (Experimental): Non-financial reward, mixed lottery, pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- N1M1P0R0 (Experimental): Non-financial reward, mixed lottery, no pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- N1M1P0R1 (Experimental): Non-financial reward, mixed lottery, no pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking
- N1L1P1R1 (Experimental): Non-financial reward, loss incentive, pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking
- N1L1P1R0 (Experimental): Non-financial reward, loss incentive, pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- N1L1P0R0 (Experimental): Non-financial reward, loss incentive, no pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- N1L1P0R1 (Experimental): Non-financial reward, loss incentive, no pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking
- F1M1P1R0 (Experimental): Financial Reward, mixed lottery, pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- F1M1P0R0 (Experimental): Financial Reward, mixed lottery, no pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- F1M1P0R1 (Experimental): Financial Reward, mixed lottery, no pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking
- F1L1P1R1 (Experimental): Financial Reward, loss incentive, pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking
- F1L1P1R0 (Experimental): Financial Reward, loss incentive, pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- F1L1P0R0 (Experimental): Financial Reward, loss incentive, no pre-commitment postcard reminders, no request physical activity advice
  Interventions: Behavioral: Walking
- F1L1P0R1 (Experimental): Financial Reward, loss incentive, no pre-commitment postcard reminders, request physical activity advice
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — Inactive Veterans will be encouraged to increase their step count to 7,000 steps per day by the end of the 12-week intervention period. Weekly the step goal will increase 15% if they were successful in reaching their goal the previous week.

SUMMARY:
Regular physical activity (PA) is essential to healthy aging. Unfortunately, only 5% of US adults meet guideline of 150 minutes of moderate exercise; Veterans and non-Veterans have similar levels of PA. A patient incentive program for PA may help. Behavioral economics suggests that the chronic inability to start and maintain a PA routine may be the result of "present bias," which is a tendency to value immediate rewards over rewards in the future. With present bias, it is always better to exercise tomorrow because the immediate gratification of watching television or surfing the internet is a more powerful motivator than the intangible and delayed benefit of future health. Patient incentives may overcome present bias by moving the rewards for exercise forward in time.

Recent randomized trials suggest that incentives for PA can be effective, but substantial gaps in knowledge prevent the implementation of a PA incentive program in Veterans Affairs (VA). First, incentive designs vary considerably. They vary by the size of the incentive, the type of incentive (cash or non-financial), the probability of earning an incentive (an assured payment for effort or a lottery-based incentive), or whether the incentive is earned after the effort is given (a gain-framed incentive) or awarded up-front and lost if the effort is not given (a loss-framed incentive). The optimal combination of these components for a Veteran population is unknown. Second, the evidence about the effective components of incentives comes from studies conducted in populations that were overwhelmingly female; often employees at large companies, with high levels of education and income. VA users, in contrast, are mostly male and lower income, and most are not employed. This is important because the investigators have theoretical reasons to believe that the effects of components of incentives are likely to vary by income and gender. Finally, few studies have managed to design an incentive such that the physical activity was maintained after the incentive was removed. Indeed, a common theme in incentivizing health behavior change is the difficulty in sustaining behavior change once the incentives are removed.

DETAILED DESCRIPTION:
The investigators propose to fill the research gaps through a Multiphase Optimization Strategy (MOST) trial of incentives for walking. A MOST trial is ideally suited for situations in which a proposed intervention has many potential intervention components. A MOST trial consists of three phases. A screening phase trial is used to efficiently identify-through a factorial designed randomized trial-the effective components of a complex intervention like incentives. A refining phase trial tests the optimal dose (size or duration) of the incentives. A confirmatory phase trial tests the optimal components and dose against a usual care control. The goal of the proposed study is to conduct the screening phase trial in 128 Veterans to identify the optimal components of incentives for increasing walking among physically inactive Veterans. All Veterans in this phase will be given various components of incentives for increasing average steps per day to 7,000 steps over a 12-week habit-building period, and then maintaining the increase through a 12-week habit maintenance period. The specific aims are:

Aim 1: Conduct a 24 factorial designed screening-phase trial of incentives for increasing average steps per day to 7,000 steps over 12 weeks among physically inactive Veterans. Every patient in the trial will be given a Fitbit Inspire activity monitor and assigned to a group that receives different components of incentives. The investigators will test four different incentive factors: 1) lottery vs. loss framed incentives, 2) financial vs. non-financial incentives, 3) a pre-commitment postcard reminder of a Veteran's stated intrinsic reason for commitment to PA vs. no pre-commitment postcard, and 4) a request for PA advice from a Veteran on staying active vs. no request. The first factor has never been tested in a population like the VA. Factors 2-4 are designed specifically to sustain the effects of incentives after the incentive is removed. Factor 4 is a novel hypothesis that has never been tested outside of educational research: specifically, that asking for advice from a Veteran is more motivating than giving advice to them, even if that Veteran is struggling with low physical activity themselves. The primary outcome is change in steps per week from baseline to week 24.

Aim 2. Conduct cost analyses and qualitative interviews. The cost of administering each component and qualitative assessments of the acceptability of each component to trial participants will inform the decision of which components to retain for the subsequent refining and confirmatory phase trials.

Aim 3. Convene an expert panel to choose components for the next phases of the MOST trial. The panel will weigh each component in terms of its effect on step counts (Aim 1), administrative costs and participant-reported qualitative assessments (Aim 2), and the strength of the theoretical basis for the component's effect on physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Veteran that receives healthcare at VA Puget Sound Health Care System
* Age 50-69
* Diagnosis of hypertension, depression or a BMI between 25-40.
* Physically inactive according to self-report. .
* 2,000-5,000 steps per day during the screening week
* Have and be able to use a smart phone.

Exclusion Criteria:

* MOVE participation in the past 4 months
* Blind
* <2,000 steps per day
* Inability to walk 20 minutes without stopping (self-report).
* Eating disorder.
* Dementia/ cognitive impairment
* Metastatic cancer, end state renal disease, hospice, palliative care, heart failure, undergoing chemotherapy, radiation or hemodialysis, have had or are on the list for an organ transplant.
* Implanted cardiovascular device such as defibrillator or ventricular device
* Active psychosis/mania/behavioral flag
* Pregnant women
* Homeless or housing insecure
* Has a paid caregiver that provides >50% of daily living activities, lives in a nursing home, assisted living facility or group home.
* Individuals that exhibit threatening, violent or inappropriate behavior during the screening phone call.
* Foot Ulcer

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Hebert, PhD BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Consent Through Baseline
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Started | 6 | 6 | 7 | 6 | 6 | 7 | 6 | 7 | 6 | 6 | 6 | 7 | 7 | 7 | 6 | 6
Completed | 3 | 5 | 3 | 1 | 3 | 4 | 2 | 0 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
Not Completed | 3 | 1 | 4 | 5 | 3 | 3 | 4 | 7 | 4 | 1 | 3 | 1 | 4 | 5 | 4 | 4
Not completed — Walked too many steps at baseline | 3 | 1 | 4 | 5 | 3 | 3 | 4 | 7 | 4 | 1 | 3 | 1 | 4 | 5 | 4 | 4
Period: Baseline to Week 12
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Started | 3 | 5 | 3 | 1 | 3 | 4 | 2 | 0 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
Completed | 3 | 4 | 3 | 1 | 3 | 3 | 2 | 0 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 12 to 24
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Started | 3 | 4 | 3 | 1 | 3 | 3 | 2 | 0 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
Completed | 2 | 4 | 2 | 1 | 3 | 3 | 2 | 0 | 2 | 4 | 3 | 6 | 3 | 1 | 1 | 2
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1 | Total
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 7 | 6 | 7 | 6 | 6 | 6 | 7 | 7 | 7 | 6 | 6 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 4 | 4 | 6 | 5 | 5 | 3 | 5 | 4 | 4 | 5 | 7 | 5 | 5 | 5 | 76
  >=65 years | 1 | 2 | 3 | 2 | 0 | 2 | 1 | 4 | 1 | 2 | 2 | 2 | 0 | 2 | 1 | 1 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (6.3) | 60.7 (5.1) | 62.3 (6.3) | 60.2 (7.8) | 60.3 (4.9) | 58.3 (6.5) | 58.3 (7.3) | 65.5 (2.6) | 58.0 (6.0) | 61.3 (6.5) | 59.0 (7.5) | 59.7 (7.1) | 61.9 (2.9) | 60.7 (3.8) | 58.3 (7.4) | 61.3 (3.9) | 60.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 3 | 1 | 2 | 2 | 1 | 3 | 1 | 0 | 2 | 23
  Male | 4 | 4 | 7 | 5 | 6 | 5 | 5 | 4 | 5 | 4 | 4 | 6 | 4 | 6 | 6 | 4 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 10
  White | 5 | 4 | 7 | 3 | 6 | 7 | 4 | 4 | 4 | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 76
  More than one race | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 7 | 6 | 6 | 7 | 6 | 7 | 6 | 6 | 6 | 7 | 7 | 7 | 6 | 6 | 102
Baseline steps [Mean (Standard Deviation); unit: steps/day] | 5358 (3185) | 4175 (690) | 4429 (2092) | 8209 (4586) | 5744 (3117) | 6740 (4100) | 6913 (3045) | 7373 (1410) | 6195 (2370) | 3456 (999) | 5193 (1683) | 4654 (1579) | 6291 (3544) | 6257 (2652) | 6313 (3544) | 7835 (5401) | 5890 (3034)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Steps Per Day From Baseline Week to Week 12
Description: The change in average steps per day from the baseline week to week 12.
Time Frame: baseline to week 12
Population: The participants in the N1L1P0R0 group were not assessed because they either walked too many or to few steps at the baseline period
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 3 | 3 | 2 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
steps/day | 4224 (719) | 4786 (6843) | 3654 (3272) | 2626 (0) | 3740 (2248) | 4493 (6036) | 3680 (96) | 4577 (97) | 1110 (1390) | 2176 (1467) | 3216 (3366) | 7002 (456) | 8158 (4016) | 3599 (226) | 2728 (0)
Statistical Analysis 1: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 12. It compares change in steps from baseline to week 12 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignment, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.418, linear mixed model; Mean Difference (Net) = -634, 90% CI 2-sided [-1924 to 655]
Statistical Analysis 2: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 12. It compares change in steps from baseline to week 12 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.033, Mixed Models Analysis; Mean Difference (Net) = -1697, 90% CI 2-sided [-3000 to -385] — Positive values represent a positive effect of lottery based rewards compared to loss-based rewards
Statistical Analysis 3: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of precommitment (PC) vs no PC factor at week 12. It compares change in steps from baseline to week 12 between subjects randomized to receive a request for PC compared to those who received no request. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.248, Mixed Models Analysis; Mean Difference (Net) = 820, 90% CI 2-sided [-347 to 1988]
Statistical Analysis 4: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no advice factor at week 12. It compares change in steps from baseline to week 12 between subjects randomized to receive a request for advice to other subjects compared to those who received no request. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.125, Mixed Models Analysis; Mean Difference (Net) = 1121, 90% CI 2-sided [82 to 2323]; Positive values represent a positive effect of requests for advice on steps compared to no request for advice

2. Secondary Outcome: Self-efficacy
Description: Measured using the Exercise Self-Efficacy Scale at baseline, week 12 and week 24 (McAuley E 1993). This scale measures self-efficacy on nine different measures from not confident (0 rating) to very confident (10 rating).The range is 0 to 10. A higher rating indicates that the respondent is more confident they will be able to overcome barriers to physical activity.
Time Frame: Measured at baseline, week 12 and 24
Population: The participants in the N1L1P0R0 group were not assessed because they walked too many steps at the baseline period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 3 | 3 | 2 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
score on a scale
  Baseline | 5.1 (1.4) | 5.7 (1.5) | 5.9 (1.4) | 2.1 (0) | 5.6 (3.7) | 5.0 (2.0) | 9.5 (0.7) | 6.4 (0.5) | 5.6 (2.9) | 5.0 (3.3) | 6.9 (1.9) | 5.9 (2.3) | 5.2 (0.2) | 4.9 (3.5) | 6.5 (2.6)
  Week 12 | 5.9 (1.1) | 6.4 (2.1) | 5.0 (2.1) | 2.1 (0) | 5.0 (1.6) | 5.6 (1.4) | 5.8 (3.1) | 6.6 (1.8) | 5.0 (1.1) | 3.2 (1.9) | 5.5 (1.0) | 6.0 (1.3) | 4.4 (1.3) | 5.6 (0) | 2.2 (1.0)
  Week 24 | 4.3 (0.2) | 6.7 (1.9) | 6.8 (2.4) | 1.3 (0) | 5.0 (1.8) | 7.1 (2.1) | 8.2 (1.7) | 4.9 (1.3) | 5.6 (1.9) | 5.0 (2.8) | 5.4 (1.5) | 6.0 (0.2) | 4.1 (0) | 4.3 (0) | 4.2 (1.3)
Statistical Analysis 1: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 12. It compares change in efficacy from baseline to week 12 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.739, Regression, Linear; Mean Difference (Net) = -0.18, 90% CI 2-sided [-1.05 to 0.70], Standard Error of Mean 0.53; Positive values represent a positive effect of financial rewards compared to non-financial rewards
Statistical Analysis 2: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 24. It compares change in efficacy from baseline to week 24 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.347, Mixed Models Analysis; Mean Difference (Net) = -0.51, 90% CI 2-sided [-1.42 to 0.39] — Positive values represent a positive effect of financial rewards compared to non-financial rewards
Statistical Analysis 3: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 12. It compares change in efficacy from baseline to week 12 between subjects randomized to receive lottery-based rewards compared to those who received loss-based rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.293, Mixed Models Analysis; Mean Difference (Net) = 0.61, 90% CI 2-sided [-0.35 to 1.57] — Positive values represent a positive effect of lottery-based rewards compared to loss-based rewards
Statistical Analysis 4: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 24. It compares efficacy at week 24 between subjects randomized to receive lottery-based rewards compared to those who received loss-based rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.599, Mixed Models Analysis; Mean Difference (Net) = 0.31, 90% CI 2-sided [-0.67 to 1.30] — Positive values represent a positive effect of lottery-based rewards compared to loss-based rewards
Statistical Analysis 5: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of precommitment (PC) vs no PC factor at week 12. It compares efficacy at week 12 between subjects randomized to receive a request for PC to other subjects compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.007, Regression, Linear; Mean Difference (Net) = 1.49, 90% CI 2-sided [0.58 to 2.40]
Statistical Analysis 6: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of precommitment (PC) vs no PC factor at week 24. It compares efficacy at week 24 between subjects randomized to receive a request for PC compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.002, Regression, Linear; Mean Difference (Net) = 1.78, 90% CI 2-sided [0.86 to 2.70]
Statistical Analysis 7: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no-advice factor at week 12. It compares efficacy at week 12 between subjects randomized to receive a request for advice to other subjects compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.068, Regression, Linear; Mean Difference (Net) = 1.02, 90% CI 2-sided [0.10 to 1.94]
Statistical Analysis 8: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no-advice factor at week 24. It compares efficacy at week 24 between subjects randomized to receive a request for advice to other subjects compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.740, Regression, Linear; Mean Difference (Net) = 0.19, 90% CI 2-sided [-0.76 to 1.14]

3. Secondary Outcome: Intrinsic/Extrinsic Motivation
Description: Measured using the Motivation for Physical Activity Measurement (MPAM) at baseline, week 12 and week 24 (Frederick CM 1993). This scale measures reasons and motivations for participating in physical activity having respondents indicate why they exercise. The scale ranges from 1=very true for me, 2= somewhat true for me, 3=neither true nor untrue for me, 4=somewhat untrue for me, 5= very untrue for me. The minimum score is 1 and the maximum is 5. Higher scores means more intrinsic motivation to exercise.
Time Frame: Measured at baseline, week 12 and 24
Population: The participants in the N1L1P0R0 group were not assessed because they walked too many steps at the baseline period
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 3 | 3 | 2 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
scores on a scale
  Baseline | 2.1 (0.7) | 2.7 (0.6) | 2.5 (0.3) | 2.8 (0) | 2.2 (0.8) | 2.6 (0.9) | 1.0 (0) | 2.0 (0.2) | 2.7 (0.4) | 1.8 (0.4) | 1.8 (0.3) | 2.1 (0.1) | 1.7 (0.2) | 1.7 (0.5) | 2.5 (2.1)
  Week 12 | 2.2 (0.3) | 2.8 (1.2) | 2.4 (0.6) | 3.0 (0) | 2.4 (0.6) | 2.1 (1.6) | 1.8 (0.1) | 1.8 (0.2) | 2.8 (0.7) | 2.0 (0.7) | 2.0 (0.4) | 2.3 (0.3) | 2.2 (0.8) | 2.0 (0) | 2.6 (2.2)
  Week 24 | 1.8 (0.5) | 2.5 (1.2) | 2.7 (0.5) | 3.0 (0) | 2.6 (0.5) | 2.4 (1.2) | 1.2 (0.2) | 2.3 (0) | 2.7 (0.8) | 1.7 (0.6) | 2.2 (0.5) | 2.1 (0.3) | 3.7 (0) | 3.7 (0) | 2.3 (1.8)
Statistical Analysis 1: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 12. It compares intrinsic motivation in week 12 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.481, Regression, Linear; Mean Difference (Net) = 0.14, 90% CI 2-sided [-0.19 to 0.47]
Statistical Analysis 2: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 24. It compares intrinsic motivation in week 24 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.388, Regression, Linear; Mean Difference (Net) = 0.18, 90% CI 2-sided [-0.16 to 0.52]
Statistical Analysis 3: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 12. It compares intrinsic motivation at week 12 between subjects randomized to receive lottery-based rewards compared to those who received loss-based rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.926, Regression, Linear; Mean Difference (Net) = -0.02, 90% CI 2-sided [-0.38 to 0.34]
Statistical Analysis 4: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 24. It compares intrinsic motivation at week 24 between subjects randomized to receive lottery-based rewards compared to those who received loss-based rewards. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.446, Regression, Linear; Mean Difference (Net) = -0.17, 90% CI 2-sided [-0.54 to 0.20]
Statistical Analysis 5: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of precommitment (PC) vs no PC factor at week 12. It compares intrinsic motivation at week 12 between subjects randomized to receive a request for PC to compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.711, Regression, Linear; Mean Difference (Net) = 0.08, 90% CI 2-sided [-0.27 to 0.42]
Statistical Analysis 6: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of precommitment (PC) vs no PC factor at week 24. It compares efficacy at week 24 between subjects randomized to receive a request for PC to compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.345, Regression, Linear; Mean Difference (Net) = -0.20, 90% CI 2-sided [-0.55 to 0.15]
Statistical Analysis 7: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no-advice factor at week 12. It compares intrinsic motivation at week 12 between subjects randomized to receive a request for advice compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.928, Regression, Linear; Mean Difference (Net) = 0.02, 90% CI 2-sided [-0.33 to 0.36]
Statistical Analysis 8: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no-advice factor at week 24. It compares intrinsic motivation at week 24 between subjects randomized to receive a request for advice to other subjects compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and survey-based outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.372, Regression, Linear; Mean Difference (Net) = -0.19, 90% CI 2-sided [-0.55 to 0.16]

4. Secondary Outcome: Mental Health
Description: Measured using the PHQ-8 depression scale at baseline, week 12 and week 24. This assessment measures depressive symptoms over the past 2 weeks. Respondents indicate how bothered they were by the following problems on a scale from 0 (not at all) to 3 (nearly every day). The minimum and maximum score are zero and 24, respectively. A lower score indicates fewer depressive symptoms.
Time Frame: Measured at baseline, week 12 and 24
Population: The participants in the N1L1P0R0 group were not assessed because they walked too many steps at the baseline period
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Number analyzed (Participants) | 3 | 4 | 3 | 1 | 3 | 3 | 2 | 2 | 5 | 3 | 6 | 3 | 2 | 2 | 2
scores on a scale
  Baseline | 4.3 (0.6) | 6.0 (6.2) | 12.7 (4.7) | 10.0 (0) | 8.3 (2.5) | 6.0 (5.3) | 4.0 (5.7) | 3.0 (1.4) | 4.4 (4.6) | 1.0 (1.4) | 4.8 (4.4) | 7.3 (7.0) | 5.0 (1.4) | 2.5 (3.5) | 3.0 (1.4)
  Week 12 | 2.0 (1.0) | 5.0 (6.7) | 15.5 (2.1) | 10.0 (0) | 5.8 (4.6) | 3.0 (0) | 9.0 (0) | 2.8 (2.5) | 6.6 (5.8) | 3.3 (2.1) | 5.3 (3.6) | 7.0 (7.2) | 3.0 (1.4) | 0 (0) | 3.5 (4.9)
  Week 24 | 2.0 (0) | 5.3 (5.3) | 7.5 (3.5) | 11 (0) | 3.3 (2.5) | 9.7 (7.4) | 7.0 (1.4) | 2.0 (2.8) | 6.0 (9.0) | 4.0 (4.0) | 7.2 (4.5) | 4.7 (6.4) | 5.0 (0) | 0 (0) | 3.5 (0.7)
Statistical Analysis 1: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P0R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 12. It compares phq8 mental health scores in week 12 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.767, Regression, Linear; Mean Difference (Net) = 0.35, 90% CI 2-sided [-1.60 to 2.3]
Statistical Analysis 2: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 24. It compares phq8 mental health scores in week 24 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.500, Regression, Linear; Mean Difference (Net) = 0.78, 90% CI 2-sided [-1.12 to 2.69]
Statistical Analysis 3: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 12. It compares phq8 mental health scores at week 12 between subjects randomized to receive lottery-based rewards compared to those who received loss-based rewards. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24, and interactions between factors and weeks; Test type: Superiority; p = 0.631, Regression, Linear; Mean Difference (Net) = 0.59, 90% CI 2-sided [-1.43 to 2.61]
Statistical Analysis 4: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 24. It compares phq8 mental health scores at week 24 between subjects randomized to receive lottery-based rewards compared to those who received loss-based rewards. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24, and interactions between factors and weeks; Test type: Superiority; p = 0.620, Regression, Linear; Mean Difference (Net) = -0.62, 90% CI 2-sided [-2.69 to 1.44]
Statistical Analysis 5: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of pre-commitment (PC) vs no PC factor at week 12. It compares phq8 mental health scores at week 12 between subjects randomized to receive a request for PC to compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.886, Regression, Linear; Mean Difference (Net) = 0.17, 90% CI 2-sided [-1.77 to 2.12]
Statistical Analysis 6: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of precommitment (PC) vs no PC factor at week 24. It compares phq8 mental health scores at week 24 between subjects randomized to receive a request for PC to compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.950, Regression, Linear; Mean Difference (Net) = -0.07, -2.03% CI 2-sided [-2.03 to 1.88]
Statistical Analysis 7: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no-advice factor at week 12. It compares phq mental health scores at week 12 between subjects randomized to receive a request for advice to other subjects compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.248, Regression, Linear; Mean Difference (Net) = -1.45, 90% CI 2-sided [-3.51 to 0.61]
Statistical Analysis 8: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no-advice factor at week 24. It compares phq mental health scores at week 24 between subjects randomized to receive a request for advice to other subjects compared to those who received no request. A linear model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, indicator for week 12 or 24 week, and interactions between factors and week indicator; Test type: Superiority; p = 0.317, Regression, Linear; Mean Difference (Net) = -1.23, 90% CI 2-sided [-3.25 to 0.79]

5. Primary Outcome: Change in Average Steps Per Day From Baseline Week to Week 24
Description: The change in average steps per day from the baseline week to week 24
Time Frame: baseline to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
Number analyzed (Participants) | 1 | 2 | 2 | 1 | 1 | 3 | 2 | 2 | 4 | 3 | 6 | 2 | 1 | 1 | 1
steps/day | 5237 (0) | 4631 (3513) | 4074 (2361) | 3804 (0) | 6414 (0) | 3844 (4122) | 2487 (3072) | 6531 (2683) | 614 (928) | 3165 (2961) | 1312 (3845) | 5939 (0) | 10675 | 4382 | 3406
Statistical Analysis 1: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of financial vs non-financial reward factor at week 24. It compares change in steps from baseline to week 24 between subjects randomized to receive financial rewards compared to those who received nonfinancial rewards. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.972, Mixed Models Analysis; Mean Difference (Net) = -35, 90% CI 2-sided [-1685 to 1616]
Statistical Analysis 2: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of lottery vs loss-framed reward factor at week 24. It compares change in steps from baseline to week 24 between subjects randomized to receive lottery-based rewards compared to those who received loss-based rewards. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Net) = -2428, 90% CI 2-sided [-4134 to -722] — Positive values represent a positive effect of lottery-based rewards compared to loss-based rewards
Statistical Analysis 3: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R1; This is the results of precommitment (PC) vs no PC factor at week 24. It compares change in steps from baseline to week 24 between subjects randomized to receive a request for PC compared to those who received no request. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.627, Mixed Models Analysis; Mean Difference (Net) = 418, 90% CI 2-sided [-999 to 1836]
Statistical Analysis 4: Comparison: F1M1P1R1 vs N1M1P1R1 vs N1M1P1R0 vs N1M1P0R0 vs N1M1P0R1 vs N1L1P1R1 vs N1L1P1R0 vs N1L1P0R1 vs F1M1P1R0 vs F1M1P0R1 vs F1L1P1R1 vs F1L1P1R0 vs F1L1P0R0 vs F1L1P0R1; This is the results of advice vs no advice factor at week 24. It compares change in steps from baseline to week 24 between subjects randomized to receive a request for advice to other subjects compared to those who received no request. A linear mixed-effect model was estimated with independent variables of demographics, steps and outcomes at baseline, indicators for each of the four factor assignments, linear week with a spline at week 12, and interactions between factors and weeks; Test type: Superiority; p = 0.842, Mixed Models Analysis; Mean Difference (Net) = 195, 90% CI 2-sided [-1417 to 1807]

ADVERSE EVENTS:
Time Frame: For 24 Weeks
Arm/Group | F1M1P1R1 | N1M1P1R1 | N1M1P1R0 | N1M1P0R0 | N1M1P0R1 | N1L1P1R1 | N1L1P1R0 | N1L1P0R0 | N1L1P0R1 | F1M1P1R0 | F1M1P0R0 | F1M1P0R1 | F1L1P1R1 | F1L1P1R0 | F1L1P0R0 | F1L1P0R1
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/7 | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic forced IRB-approved changes to recruitment procedures to obviate in-person recruitment. Recruitment was slowed dramatically and we missed our target enrollment. All statistical tests are underpowered.

Because of slow delivery of mailed study material, we received IRB approval to randomize patients at consent rather than after the week-long baseline period. This resulted in random imbalance in assignment to treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT04518943/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT04518943/ICF_000.pdf